CLINICAL TRIAL: NCT00136370
Title: Preventing Serious Neonatal and Maternal Peripartum Infections in Developing Country Settings With a High Prevalence of HIV Infection: Assessment of the Disease Burden and Evaluation of an Affordable Intervention in Soweto, South Africa
Brief Title: Prevention of Perinatal Sepsis (PoPS): Evaluation of Chlorhexidine Wipes of Birth Canal and Newborn
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Bill and Melinda Gates Foundation (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); National Vaccine Program Office (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCID-3842; #U50 CCU021960, 02075; RFA CI05-059
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Infant, Newborn, Diseases; Sepsis; Puerperal Infection
Keywords: Chlorhexidine; Prevention; Neonatal sepsis; Peripartum infections
MeSH Terms: conditions — Infant, Newborn, Diseases; Sepsis; Puerperal Infection; Neonatal Sepsis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Chlorhexidine Vaginal Wipe
  Interventions: Drug: Chlorhexidine; Procedure: Birth canal wipe
- 2 (Placebo Comparator): Sterile water external genital wipe
  Interventions: Procedure: sterile water external genital wipe

INTERVENTIONS:
Drug: Chlorhexidine
  Arms: 1
Procedure: Birth canal wipe
  Arms: 1
Procedure: sterile water external genital wipe
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether use of the disinfectant chlorhexidine administered to the birth canal during labour and newborn at delivery can protect a woman and her baby from bacterial infections after birth. If effective, this could be used as an inexpensive alternative to antibiotics to prevent newborn infections in resource-poor countries.

DETAILED DESCRIPTION:
We are conducting a randomized, controlled clinical trial in Soweto, South Africa to evaluate the efficacy of 0.5% chlorhexidine wipes of the birth canal during labour and of the infant at birth in reducing 1) vertical transmission of leading pathogenic bacteria from mother to child during labour and delivery, and 2) incidence of neonatal sepsis and maternal peripartum infection, in comparison to external genitalia sterile water wipes. In conjunction with this, we will compare vaginal carriage of bacteria commonly associated with neonatal sepsis and maternal peripartum infection among HIV-infected and non-infected pregnant women who deliver at the only public hospital in Soweto, and will characterize the burden of disease and risk factors for maternal peripartum infection and serious neonatal infections in this population by conducting active prospective surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Plan to deliver at Chris Hani Baragwanath Hospital or one of its satellite clinics
* Plan to remain in Soweto for at least two months after delivery
* Are able to understand and give informed consent
* Are at least 15 years old at time of registration

Exclusion Criteria:

* Planned delivery by caesarean section
* Antenatal ultrasound revealing major fetal congenital anomalies
* Have known or suspected condition in which vaginal exams are contraindicated, e.g. placenta previa
* Have a history of allergic reaction to any topical antiseptic solution
* Present to labour ward with infant born before arrival
* Present to labour ward with significant vaginal bleeding during labour
* Present with known intrauterine fetal death prior to randomization
* Subject noted to be in full cervical dilatation or have baby's head on perineum
* Infant noted to be in face presentation on first vaginal examination
* Noted to have genital ulcers present on first vaginal examination

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2004-04; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Rates of culture-confirmed or clinical neonatal sepsis, < 3 days of life
Rate of vertical transmission of colonization with group B streptococcus (GBS)

SECONDARY OUTCOMES:
Rates of culture-confirmed or clinical neonatal sepsis (non-nosocomial), 3 to 28 days of life
Rates of serious maternal per partum infections including: endometritis, culture-confirmed post-partum sepsis, and post-partum perineal wound infection
Rates of neonatal hospitalization, < 3 days of life
Rates of neonatal hospitalization, < 28 days of life
Rates of neonatal hospitalization, suspected sepsis
Rate of vertical transmission of colonization with E. coli or Klebsiella species

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Schrag, DPhil, Principal Investigator — Centers for Disease Control and Prevention; Shabir Madhi, MD, PhD, Principal Investigator — Respiratory and Meningeal Pathogens Research Unit
Locations (1):
- Chris Hani Baragwanath Hospital, Soweto, Gauteng, South Africa

REFERENCES:
- [Background] Christensen KK, Christensen P, Dykes AK, Kahlmeter G. Chlorhexidine for prevention of neonatal colonization with group B streptococci. III. Effect of vaginal washing with chlorhexidine before rupture of the membranes. Eur J Obstet Gynecol Reprod Biol. 1985 Apr;19(4):231-6. doi: 10.1016/0028-2243(85)90034-6. PMID 3891445
- [Background] Taha TE, Biggar RJ, Broadhead RL, Mtimavalye LA, Justesen AB, Liomba GN, Chiphangwi JD, Miotti PG. Effect of cleansing the birth canal with antiseptic solution on maternal and newborn morbidity and mortality in Malawi: clinical trial. BMJ. 1997 Jul 26;315(7102):216-9; discussion 220. doi: 10.1136/bmj.315.7102.216. PMID 9253269
- [Background] Kollee LA, Speyer I, van Kuijck MA, Koopman R, Dony JM, Bakker JH, Wintermans RG. Prevention of group B streptococci transmission during delivery by vaginal application of chlorhexidine gel. Eur J Obstet Gynecol Reprod Biol. 1989 Apr;31(1):47-51. doi: 10.1016/0028-2243(89)90025-7. PMID 2653894
- [Background] Burman LG, Christensen P, Christensen K, Fryklund B, Helgesson AM, Svenningsen NW, Tullus K. Prevention of excess neonatal morbidity associated with group B streptococci by vaginal chlorhexidine disinfection during labour. The Swedish Chlorhexidine Study Group. Lancet. 1992 Jul 11;340(8811):65-9. doi: 10.1016/0140-6736(92)90393-h. PMID 1352011
- [Background] Adriaanse AH, Kollee LA, Muytjens HL, Nijhuis JG, de Haan AF, Eskes TK. Randomized study of vaginal chlorhexidine disinfection during labor to prevent vertical transmission of group B streptococci. Eur J Obstet Gynecol Reprod Biol. 1995 Aug;61(2):135-41. doi: 10.1016/0301-2115(95)02134-s. PMID 7556834
- [Background] Rouse DJ, Hauth JC, Andrews WW, Mills BB, Maher JE. Chlorhexidine vaginal irrigation for the prevention of peripartal infection: a placebo-controlled randomized clinical trial. Am J Obstet Gynecol. 1997 Mar;176(3):617-22. doi: 10.1016/s0002-9378(97)70557-x. PMID 9077616
- [Background] Stray-Pedersen B, Bergan T, Hafstad A, Normann E, Grogaard J, Vangdal M. Vaginal disinfection with chlorhexidine during childbirth. Int J Antimicrob Agents. 1999 Aug;12(3):245-51. doi: 10.1016/s0924-8579(99)00068-0. PMID 10461843
- [Background] Facchinetti F, Piccinini F, Mordini B, Volpe A. Chlorhexidine vaginal flushings versus systemic ampicillin in the prevention of vertical transmission of neonatal group B streptococcus, at term. J Matern Fetal Neonatal Med. 2002 Feb;11(2):84-8. doi: 10.1080/jmf.11.2.84.88. PMID 12375548
- [Derived] Cutland CL, Schrag SJ, Zell ER, Kuwanda L, Buchmann E, Velaphi SC, Groome MJ, Adrian PV, Madhi SA; PoPS trial team. Maternal HIV infection and vertical transmission of pathogenic bacteria. Pediatrics. 2012 Sep;130(3):e581-90. doi: 10.1542/peds.2011-1548. Epub 2012 Aug 6. PMID 22869824
- [Derived] Schrag SJ, Cutland CL, Zell ER, Kuwanda L, Buchmann EJ, Velaphi SC, Groome MJ, Madhi SA; PoPS Trial Team. Risk factors for neonatal sepsis and perinatal death among infants enrolled in the prevention of perinatal sepsis trial, Soweto, South Africa. Pediatr Infect Dis J. 2012 Aug;31(8):821-6. doi: 10.1097/INF.0b013e31825c4b5a. PMID 22565291
- [Derived] Cutland CL, Madhi SA, Zell ER, Kuwanda L, Laque M, Groome M, Gorwitz R, Thigpen MC, Patel R, Velaphi SC, Adrian P, Klugman K, Schuchat A, Schrag SJ; PoPS Trial Team. Chlorhexidine maternal-vaginal and neonate body wipes in sepsis and vertical transmission of pathogenic bacteria in South Africa: a randomised, controlled trial. Lancet. 2009 Dec 5;374(9705):1909-16. doi: 10.1016/S0140-6736(09)61339-8. Epub 2009 Oct 19. PMID 19846212